CLINICAL TRIAL: NCT00861094
Title: Phase II-III Study Comparing Radiochemotherapy With the FOLFOX Regimen Versus Radiochemotherapy With 5FU-cisplatin (Herskovic Regimen) in First Line Treatment of Patients With Inoperable Oesophageal Cancer.
Brief Title: Radiation Therapy + Combination Chemotherapy as 1st-Line Therapy for Patients With Inoperable Esophageal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595050; FRE-FNCLCC- ACCORD-17-0707; EU-20848
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Oxaliplatin; Radiotherapy; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX and radiotherapy (Experimental): Oxaliplatin (85mg/m2); Folinic Acid (200mg/m2); 5-FU (400mg/m2-Bolus and 1600mg/m2 over 46h)- once every two weeks for six cycles
  Interventions: Drug: 5-FU; Drug: oxaliplatin; Radiation: radiation therapy; Drug: Folinic Acid
- 5-FU / cisplatin and radiotherapy (Experimental): 5-FU (100mg/m2); Cisplatin (75mg/m2)
  Interventions: Drug: cisplatin; Drug: 5-FU; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
  Arms: 5-FU / cisplatin and radiotherapy
Drug: 5-FU
  Other Names: 5-Fluorouracil
Drug: oxaliplatin
  Arms: FOLFOX and radiotherapy
Radiation: radiation therapy
Drug: Folinic Acid
  Arms: FOLFOX and radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, leucovorin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This randomized phase II/III trial is studying radiation therapy and two different combination chemotherapy regimens to compare how well they work as first-line therapy in treating patients with esophageal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of radiochemotherapy comprising oxaliplatin, fluorouracil, and leucovorin calcium (FOLFOX regimen) vs fluorouracil and cisplatin (Herskovic regimen) in patients with inoperable esophageal cancer. (Phase II)
* To assess the endoscopic complete response rate in patients treated with these regimens. (Phase II)
* To compare the event-free survival of patients treated with these regimens. (Phase III)

Secondary

* To assess the toxicity profile of these regimens using the NCI CTC v2.0 criteria. (Phase II)
* To compare the overall survival, endoscopic complete response rate, incidence of grade 3-4 toxicities, and time to treatment failure in patients treated with these regimens. (Phase III)
* To evaluate the quality of life of these patients using EORTC QLQ-C30 (version 3) and a validated disease-specific module EORTC QLQ-OES18. (Phase III)

OUTLINE: This is a multicenter study. Patients are stratified according to histological type (adenocarcinoma or adenosquamous carcinoma vs squamous cell carcinoma), pretreatment weight loss within the past 6 months (grade 1 [< 10%] vs grade 2 [≥ 10%]), ECOG performance status (0 vs 1 vs 2), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (modified FOLFOX 4 regimen): Patients undergo radiotherapy 5 days a week for 5 weeks. Beginning concurrently with radiotherapy, patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment with chemotherapy repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (Herskovic regimen): Patients undergo radiotherapy as in arm I. Patients also receive cisplatin IV continuously over 24 hours on day 1 and fluorouracil IV continuously over 96 hours on days 1-4 of weeks 1, 5, 8, and 11 in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, periodically during study therapy, and then every 6 months for 1 year and annually for 3 years after completion of study therapy.

After completion of study therapy, patients are followed at 4 weeks and then every 3-6 months until disease progression.

PROJECTED ACCRUAL: A total of 97 patients will be accrued for the phase II portion of the study. A total of 169 patients will be accrued for the phase III portion of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma, squamous cell carcinoma, or adenosquamous carcinoma of the esophagus

  * Locally advanced disease (any T, N0 or N1, M0 or M1a)

    * No metastatic disease, except for tumor involvement of the upper third of the esophagus or cervical esophageal tumor with regional nodes, or tumor involvement of the lower third of the esophagus with celiac nodes (M1a)

      * Cervical primary tumor with positive supraclavicular or cervical lymph nodes (defined as N1) allowed
      * No radiographic evidence of enlarged (≥ 1.5 cm) celiac lymph nodes by CT scan or echography
  * No small cell or undifferentiated carcinoma of the esophagus
  * No multiple carcinomas of the esophagus (i.e., > 1 esophageal tumor)
  * No cardia tumor (Siewert II) or gastric tumor extension to the esophagus (Siewert III)

    * Esophageal tumor extension to the cardia (Siewert I) (center of the tumor lying > 1 cm-5 cm above gastroesophageal junction) allowed
* Inoperable disease OR surgery is contraindicated
* No tracheo-esophageal fistula or invasion of the tracheo-bronchial tree

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Creatinine < 15 mg/L
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 2.5 times ULN
* Prothrombin time ≥ 60%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Caloric intake sufficient (i.e., > 1,000 Kcal/m²/day) (orally or with gastrostomy)
* No weight loss > 20% normal body weight within the past 3 months
* No complete dysphagia
* No exclusive requirement for parenteral nutrition
* No peripheral neuropathy > grade 1

  * No sensitive peripheral neuropathy with functional impairment
* No auditory disorders
* No other prior malignancies except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix or stage I or II node-negative head and neck cancer that was curatively treated > 3 years ago
* No myocardial infarction within the past 6 months

  * Patients who have had a myocardial infarction > 6 months ago are eligible provided there is no transient ischemia by thallium myocardial scintigraphy and patient is able to undergo chemotherapy , as determined by a cardiologist
* No other serious illness or medical condition (e.g., symptomatic coronary disease, left ventricular failure, or uncontrolled infection)
* No stage II-IV arterial disease, according to the DE LERICHE and FONTAINE classification
* No geographical, social, or psychological circumstances preventing regular follow-up

PRIOR CONCURRENT THERAPY:

* No prior treatment for esophageal cancer (e.g., surgery, chemotherapy, or radiotherapy)
* No prior cervical, thoracic, or abdominal radiotherapy with field overlapping the proposed esophageal radiotherapy field
* More than 30 days since prior experimental drugs or participation in another clinical trial
* No other concurrent anticancer therapy
* No concurrent phenytoin or yellow fever vaccine
* No concurrent high-dose, long-term corticosteroids
* No concurrent calcium gluconate/magnesium sulfate infusions
* No concurrent hematopoietic growth factors
* No concurrent esophageal dilatation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who complete the full study treatment (Phase II) | 12 weeks
Endoscopic complete response rate (Phase II) | 12 weeks
Progression-free survival (Phase III) | Until progression

SECONDARY OUTCOMES:
Safety profile as assessed by NCI CTC v2.0 (Phase II) | Total duration of the trial
Overall survival (Phase III) | Total duration of the trial
Complete response rate (Phase III) | Total duration of the trial
Time to treatment failure (Phase III) | Total duration of the trial
Incidence of grade 3-4 toxicities (Phase III) | Total duration of the trial
Quality of life as assessed by EORTC QLQ-C30 (version 3) and EORTC QLQ-OES18 (Phase III) | Total duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Conroy, MD, Principal Investigator — Centre Alexis Vautrin
Locations (28):
- France (28):
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Polyclinique Du Parc, Caen
  - Centre Regional Francois Baclesse, Caen
  - Hopital Du Bocage, Dijon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Tenon, Paris
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - CHU - Robert Debre, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Clinique Du Parc, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Winter A, Cuer B, Conroy T, Juzyna B, Gourgou S, Mollevi C, Touraine C. Flexible modeling of longitudinal health-related quality of life data accounting for informative dropout in a cancer clinical trial. Qual Life Res. 2023 Mar;32(3):669-679. doi: 10.1007/s11136-022-03252-6. Epub 2022 Sep 17. PMID 36115002
- [Derived] Cuer B, Conroy T, Juzyna B, Gourgou S, Mollevi C, Touraine C. Joint modelling with competing risks of dropout for longitudinal analysis of health-related quality of life in cancer clinical trials. Qual Life Res. 2022 May;31(5):1359-1370. doi: 10.1007/s11136-021-03040-8. Epub 2021 Nov 24. PMID 34817733
- [Derived] Cuer B, Mollevi C, Anota A, Charton E, Juzyna B, Conroy T, Touraine C. Handling informative dropout in longitudinal analysis of health-related quality of life: application of three approaches to data from the esophageal cancer clinical trial PRODIGE 5/ACCORD 17. BMC Med Res Methodol. 2020 Sep 3;20(1):223. doi: 10.1186/s12874-020-01104-w. PMID 32883216
- [Derived] Conroy T, Galais MP, Raoul JL, Bouche O, Gourgou-Bourgade S, Douillard JY, Etienne PL, Boige V, Martel-Lafay I, Michel P, Llacer-Moscardo C, Francois E, Crehange G, Abdelghani MB, Juzyna B, Bedenne L, Adenis A; Federation Francophone de Cancerologie Digestive and UNICANCER-GI Group. Definitive chemoradiotherapy with FOLFOX versus fluorouracil and cisplatin in patients with oesophageal cancer (PRODIGE5/ACCORD17): final results of a randomised, phase 2/3 trial. Lancet Oncol. 2014 Mar;15(3):305-14. doi: 10.1016/S1470-2045(14)70028-2. Epub 2014 Feb 18. PMID 24556041